CLINICAL TRIAL: NCT06222528
Title: Brief Personalized Videos to Reduce Stigma and Increase Treatment-seeking Behavior Among Adolescents With Depression
Brief Title: Reducing Stigma and Increasing Treatment Seeking Intentions Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Doron Amsalem, Assistant Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8317
Record Dates: First submitted 2024-01-16; First posted 2024-01-24 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Stigma, Social; Mental Health Disorder; Adolescent Behavior; Depression
MeSH Terms: conditions — Social Stigma; Mental Disorders; Adolescent Behavior; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Brief video intervention (Black Girl) (Experimental): A brief social contact-based video with a Black girl protagonist
  Interventions: Behavioral: Brief video intervention (Black Girl)
- Brief video intervention (Black Boy) (Experimental): A brief social contact-based video with a Black boy protagonist
  Interventions: Behavioral: Brief video intervention (Black Boy)
- Brief video intervention (Latinx Girl) (Experimental): A brief social contact-based video with a Latinx girl protagonist
  Interventions: Behavioral: Brief video intervention (Latinx Girl)
- Brief video intervention (Latinx Boy) (Experimental): A brief social contact-based video with a Latinx boy protagonist
  Interventions: Behavioral: Brief video intervention (Latinx Boy)
- Brief video intervention (White Girl) (Experimental): A brief social contact-based video with a White girl protagonist
  Interventions: Behavioral: Brief video intervention (White Girl)
- Brief video intervention (White Boy) (Experimental): A brief social contact-based video with a White boy protagonist
  Interventions: Behavioral: Brief video intervention (White Boy)
- Brief video intervention (Nonbinary or transgender) (Experimental): A brief social contact-based video with a nonbinary or transgender protagonist
  Interventions: Behavioral: Brief video intervention (Nonbinary or transgender)
- Control (Active Comparator): A brief video control condition with psychoeducation on depression and help seeking
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Brief video intervention (Black Girl) — A brief social contact-based video. The video presented a young Black girl, a professional actor, sharing her scripted personal story of struggles with depression and raising themes of recovery and hope.
  Arms: Brief video intervention (Black Girl)
Behavioral: Brief video intervention (Black Boy) — A brief social contact-based video. The video presented a young Black boy, a professional actor, sharing his scripted personal story of struggles with depression and raising themes of recovery and hope.
  Arms: Brief video intervention (Black Boy)
Behavioral: Brief video intervention (Latinx Girl) — A brief social contact-based video. The video presented a young Latinx girl, a professional actor, sharing her scripted personal story of struggles with depression and raising themes of recovery and hope.
  Arms: Brief video intervention (Latinx Girl)
Behavioral: Brief video intervention (Latinx Boy) — A brief social contact-based video. The video presented a young Latinx boy, a professional actor, sharing his scripted personal story of struggles with depression and raising themes of recovery and hope.
  Arms: Brief video intervention (Latinx Boy)
Behavioral: Brief video intervention (White Girl) — A brief social contact-based video. The video presented a young White girl, a professional actor, sharing her scripted personal story of struggles with depression and raising themes of recovery and hope.
  Arms: Brief video intervention (White Girl)
Behavioral: Brief video intervention (White Boy) — A brief social contact-based video. The video presented a young White boy, a professional actor, sharing his scripted personal story of struggles with depression and raising themes of recovery and hope.
  Arms: Brief video intervention (White Boy)
Behavioral: Brief video intervention (Nonbinary or transgender) — A brief social contact-based video. The video presented a young nonbinary or transgender adolescent, a professional actor, sharing their scripted personal story of struggles with depression and raising themes of recovery and hope.
  Arms: Brief video intervention (Nonbinary or transgender)
Behavioral: Control Condition — A video that will provide information about depression and how to seek help but does not include a personal story.
  Arms: Control

SUMMARY:
Depression is a leading cause of illness and disability in teenagers. Longer duration of untreated depression (DUD) is associated with greater severity, poorer outcome, and cognitive impairment. Stigma toward people with depression has been identified as a barrier to seeking help; therefore, reducing stigma toward young people at depressive risk could enhance their receptivity to seeking treatment. Social contact is a form of interpersonal contact with members of the stigmatized group and the most effective type of intervention for improvement in stigma-related knowledge and attitudes.

In a prior study, the investigators developed short video interventions to reduce stigma and increase treatment seeking among adolescents with depression. The videos feature adolescent protagonists varied by race/ethncitiy and gender (Black girl, Black boy, White girl, White boy, Hispanic girl, Hispanic boy, nonbinary or transgender adolescent) who will share their experiences with depression, challenges, and recovery process. The investigators would like to conduct a randomized controlled trial (RCT) to test the efficacy of these tailored videos as compared to a video control condition (which provides information about depression and how to seek help but does not include a personal story) on reducing self-stigma and increasing help-seeking intentions and behavior at baseline, post, 2 week follow-up, and 4 week follow-up among adolescents ages 14-18 recruited via Cloudresearch. The videos will be shown again at 2 week follow-up.

DETAILED DESCRIPTION:
In a randomized control trial (RCT) with pre-, post-intervention, and 2 and 4 week follow-up assessments, the investigators aim to test the efficacy of brief social contact video interventions, varying protagonist race/ethnicity, as compared to video control in reducing depression related stigma and increasing treatment-seeking intentions and behavior among adolescents ages 14-18 recruited via Cloudresearch, a crowdsourcing platform. The control condition will include a video that will provide information about depression and how to seek help but does not include a personal story. The tailored video interventions will be assigned based on participant demographics and will include adolescent protagonists varied by race/ethnicity and gender (Black girl, Black boy, White girl, White boy, Hispanic girl, Hispanic boy, nonbinary or transgender adolescent). Videos will be shown at baseline and 2 week follow-up. The investigators hypothesize that 1) Brief social contact-based video interventions will reduce stigma towards depression and increase treatment-seeking intentions and behavior compared to video control which provides information about depression and help seeking but does not include a personal story.

ELIGIBILITY:
Inclusion Criteria:

* Ages 14-18
* English speaking
* US Residents

Exclusion Criteria:

* Age less than 14 or greater than 18
* Non-English speaking
* Non-US Resident

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1200 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-08-17 (Actual); Study Completion 2024-08-17 (Actual)

PRIMARY OUTCOMES:
Depression Stigma | Baseline
  The Depression Stigma Scale (DSS) is a self-report scale comprised of two 9-item subscales measuring participants' personal beliefs about depression and participants' beliefs about others' attitudes (Griffiths et al., 2004). The current study will only utilize the personal beliefs subscale. Each item is rated on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). Scores range from 9 to 45. Higher scores indicate more stigma.
Depression Stigma | Post (immediately after the videos are shown)
  The Depression Stigma Scale (DSS) is a self-report scale comprised of two 9-item subscales measuring participants' personal beliefs about depression and participants' beliefs about others' attitudes (Griffiths et al., 2004). The current study will only utilize the personal beliefs subscale. Each item is rated on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). Scores range from 9 to 45. Higher scores indicate more stigma.
Depression Stigma | 2 week follow-up
  The Depression Stigma Scale (DSS) is a self-report scale comprised of two 9-item subscales measuring participants' personal beliefs about depression and participants' beliefs about others' attitudes (Griffiths et al., 2004). The current study will only utilize the personal beliefs subscale. Each item is rated on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). Scores range from 9 to 45. Higher scores indicate more stigma.
Depression Stigma | 4 week follow-up
  The Depression Stigma Scale (DSS) is a self-report scale comprised of two 9-item subscales measuring participants' personal beliefs about depression and participants' beliefs about others' attitudes (Griffiths et al., 2004). The current study will only utilize the personal beliefs subscale. Each item is rated on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). Scores range from 9 to 45. Higher scores indicate more stigma.
Attitude Towards Seeking Professional Psychological Help | Baseline
  Treatment seeking intentions will be measured using three items from the Attitudes Towards Seeking Professional Psychological Help Scale (ATSPPHS) Scale (Elhai et al., 2008). Items include: 'I might want to have psychological counselling in the future', 'I would want to get psychological help if I were worried or upset for a long period of time' and 'A person with an emotional problem is not likely to solve it alone; he or she is more likely to solve it with professional help'. Responses range from 1 (disagree) to 4 (agree). Total scores range from 3 to 12 with higher scores indicating higher treatment seeking intentions.
Attitude Towards Seeking Professional Psychological Help | Post (immediately after the videos are shown)
  Treatment seeking intentions will be measured using three items from the Attitudes Towards Seeking Professional Psychological Help Scale (ATSPPHS) Scale (Elhai et al., 2008). Items include: 'I might want to have psychological counselling in the future', 'I would want to get psychological help if I were worried or upset for a long period of time' and 'A person with an emotional problem is not likely to solve it alone; he or she is more likely to solve it with professional help'. Responses range from 1 (disagree) to 4 (agree). Total scores range from 3 to 12 with higher scores indicating higher treatment seeking intentions.
Attitude Towards Seeking Professional Psychological Help | 2 week follow-up
  Treatment seeking intentions will be measured using three items from the Attitudes Towards Seeking Professional Psychological Help Scale (ATSPPHS) Scale (Elhai et al., 2008). Items include: 'I might want to have psychological counselling in the future', 'I would want to get psychological help if I were worried or upset for a long period of time' and 'A person with an emotional problem is not likely to solve it alone; he or she is more likely to solve it with professional help'. Responses range from 1 (disagree) to 4 (agree). Total scores range from 3 to 12 with higher scores indicating higher treatment seeking intentions.
Attitude Towards Seeking Professional Psychological Help | 4 week follow-up
  Treatment seeking intentions will be measured using three items from the Attitudes Towards Seeking Professional Psychological Help Scale (ATSPPHS) Scale (Elhai et al., 2008). Items include: 'I might want to have psychological counselling in the future', 'I would want to get psychological help if I were worried or upset for a long period of time' and 'A person with an emotional problem is not likely to solve it alone; he or she is more likely to solve it with professional help'. Responses range from 1 (disagree) to 4 (agree). Total scores range from 3 to 12 with higher scores indicating higher treatment seeking intentions.

SECONDARY OUTCOMES:
Emotional engagement | Post (immediately after the videos are shown
  Emotional engagement will be measured using the Emotional Engagement Scale (de Vreede et al., 2019). The scale includes three items asking about emotional engagement (e.g., "I care about the contents of this video"), and response choices range from 1 (strongly disagree) to 4 (strongly agree). Total scores range from 3 to 12, with higher scores indicating greater emotional engagement.
Emotional engagement | 2 week follow-up
  Emotional engagement will be measured using the Emotional Engagement Scale (de Vreede et al., 2019). The scale includes three items asking about emotional engagement (e.g., "I care about the contents of this video"), and response choices range from 1 (strongly disagree) to 4 (strongly agree). Total scores range from 3 to 12, with higher scores indicating greater emotional engagement.
Treatment related stigma | Baseline
  Treatment-related stigma will be measured with the Self-Stigma of Seeking Help scale (SSOSH-3) (Brenner et al., 2021). Items include "I would feel inadequate if I went to a therapist for psychological help," "It would make me feel inferior to ask a therapist for help," and "If I went to a therapist, I would be less satisfied with myself." Response range from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 3 to 15, with higher scores indicating greater stigma.
Treatment related stigma | Post (immediately after the videos are shown)
  Treatment-related stigma will be measured with the Self-Stigma of Seeking Help scale (SSOSH-3) (Brenner et al., 2021). Items include "I would feel inadequate if I went to a therapist for psychological help," "It would make me feel inferior to ask a therapist for help," and "If I went to a therapist, I would be less satisfied with myself." Response range from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 3 to 15, with higher scores indicating greater stigma.
Treatment related stigma | 2 week follow-up
  Treatment-related stigma will be measured with the Self-Stigma of Seeking Help scale (SSOSH-3) (Brenner et al., 2021). Items include "I would feel inadequate if I went to a therapist for psychological help," "It would make me feel inferior to ask a therapist for help," and "If I went to a therapist, I would be less satisfied with myself." Response range from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 3 to 15, with higher scores indicating greater stigma.
Treatment related stigma | 4 week follow-up
  Treatment-related stigma will be measured with the Self-Stigma of Seeking Help scale (SSOSH-3) (Brenner et al., 2021). Items include "I would feel inadequate if I went to a therapist for psychological help," "It would make me feel inferior to ask a therapist for help," and "If I went to a therapist, I would be less satisfied with myself." Response range from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 3 to 15, with higher scores indicating greater stigma.
Barriers to Access to Care Evaluation (BACE V3) | Baseline
  Barriers to care will be measured with items selected from the Barriers to Access to Care Evaluation (BACE v3) (Clement et al., 2012). Response range from 0 (not at all) to 3 (a lot). Total scores range from 0 to 24, with higher scores indicating greater barriers.
Barriers to Access to Care Evaluation (BACE V3) | Post (immediately after the videos are shown)
  Barriers to care will be measured with items selected from the Barriers to Access to Care Evaluation (BACE v3) (Clement et al., 2012). Response range from 0 (not at all) to 3 (a lot). Total scores range from 0 to 24, with higher scores indicating greater barriers.
Barriers to Access to Care Evaluation (BACE V3) | 2 week follow-up
  Barriers to care will be measured with items selected from the Barriers to Access to Care Evaluation (BACE v3) (Clement et al., 2012). Response range from 0 (not at all) to 3 (a lot). Total scores range from 0 to 24, with higher scores indicating greater barriers.
Barriers to Access to Care Evaluation (BACE V3) | 4 week follow-up
  Barriers to care will be measured with items selected from the Barriers to Access to Care Evaluation (BACE v3) (Clement et al., 2012). Response range from 0 (not at all) to 3 (a lot). Total scores range from 0 to 24, with higher scores indicating greater barriers.
Mental Health Treatment | Baseline
  One item will be utilized to measure prior mental health treatment: Have you ever received mental health treatment?
Actual help seeking | 2 week follow-up
  Two items will be utilized to measure help seeking: Over the past 2 weeks, have you sought out mental health treatment? and Over the past 2 weeks, did you feel more able/willing to open up to others about how you are feeling?
Actual help seeking | 4 week follow-up
  Two items will be utilized to measure help seeking: Over the past 4 weeks, have you sought out mental health treatment? and Over the past 4 weeks, did you feel more able/willing to open up to others about how you are feeling?

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griffiths KM, Christensen H, Jorm AF, Evans K, Groves C. Effect of web-based depression literacy and cognitive-behavioural therapy interventions on stigmatising attitudes to depression: randomised controlled trial. Br J Psychiatry. 2004 Oct;185:342-9. doi: 10.1192/bjp.185.4.342. PMID 15458995
- [Background] Elhai JD, Schweinle W, Anderson SM. Reliability and validity of the Attitudes Toward Seeking Professional Psychological Help Scale-Short Form. Psychiatry Res. 2008 Jun 30;159(3):320-9. doi: 10.1016/j.psychres.2007.04.020. Epub 2008 Apr 22. PMID 18433879
- [Background] de Vreede T, Andel SA, de Vreede GJ, Spector P, Singh V, Padmanabhan B. What is engagement and how do we measure it? Toward a domain independent definition and scale. Proceedings of the 52nd Hawaii International Conference on System Sciences. 2019, Hawaii. p. 749-758.
- [Background] Clement S, Brohan E, Jeffery D, Henderson C, Hatch SL, Thornicroft G. Development and psychometric properties the Barriers to Access to Care Evaluation scale (BACE) related to people with mental ill health. BMC Psychiatry. 2012 Jun 20;12:36. doi: 10.1186/1471-244X-12-36. PMID 22546012
- [Background] Brenner RE, Colvin KF, Hammer JH, Vogel DL. Using Item Response Theory to Develop Revised (SSOSH-7) and Ultra-Brief (SSOSH-3) Self-Stigma of Seeking Help Scales. Assessment. 2021 Jul;28(5):1488-1499. doi: 10.1177/1073191120958496. Epub 2020 Sep 25. PMID 32975438